CLINICAL TRIAL: NCT01639794
Title: An Irish Observational Study to Evaluate LUTS Storage Symptom Improvement in Men Being Treated With Vesitirim™ (Solifenacin)
Brief Title: Vesitirim™ in Men Postmarketing Observational Study
Acronym: VIM
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: VES-IE-001
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Lower Urinary Tract Symptoms (LUTS); Overactive Bladder (OAB)
Keywords: LUTS (Lower Urinary Tract Symptoms); Overactive Bladder (OAB)Vesitirim; Solifenacin; Anti-muscarinic treatment; Cholinergic receptor antagonist; Storage Symptom improvement
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Male patients with non-neurogenic LUTS taking VESITRIM: Male patients diagnosed with non-neurogenic Lower Urinary Tract Symptoms (LUTS) with bothersome storage disorder defined as urgency, and/or frequency and/or Urgency Urinary Incontinence (UUI)
  Interventions: Drug: Vesitirim™ (Solifenacin)

INTERVENTIONS:
Drug: Vesitirim™ (Solifenacin) — Oral
  Other Names: Solifenacin

SUMMARY:
This is an observational study which will look at the improvement in Lower Urinary Tract Symptoms (LUTS) in Irish men being treated with Vesitirim™ (solifenacin).

Vesitirim™ is a competitive specific muscarinic receptor antagonist and has been used extensively for the treatment of OAB (Over Active Bladder) in women and has shown significant impact on urgency, frequency and incontinence in females. It is also indicated for the symptomatic treatment of urgency incontinence and/or increased urinary frequency and urgency in men. The purpose of this study is to evaluate LUTS storage symptom improvement in men with non neurogenic LUTS who have been prescribed Vesitirim™.

The effect of Vesitirim (solifenacin) treatment on bothersome symptoms improvement will be measured using Over Active Bladder-q Short Form (OAB-qSF) and the Perception of Treatment Satisfaction (TS-VAS). The study will also help define some of the characteristics of the male population in Ireland who are treated with Vesitirim™ (solifenacin) as well as evaluating the effect of Vesitirim™ monotherapy or combination therapy on storage symptoms improvement (urgency, frequency and urge incontinence) using a bladder diary and IPSS (International Prostate Symptom Score). The study will also evaluate the effect of Vesitirim™ monotherapy or combination therapy on nocturia using IPSS. The impact of LUTS on quality of life will also be assessed. Data will also be collected regarding adverse drug reactions.

DETAILED DESCRIPTION:
This is a post marketing, non-interventional study (NIS) of patients who are to be treated with Vesitirim™. The decision whether or not to treat with Vesitirim™ will be made by the treating physician prior to the entry of the patient into the study. The patient will be informed of the study and written consent will be obtained prior to screening and determination of eligibility.

No study drug will be supplied as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-neurogenic Lower Urinary Tract Symptoms (LUTS) with bothersome storage disorder defined as urgency, and/or frequency and/or Urge Urinary Incontinence (UUI) at the discretion of the Investigator
* Eligible to start Vesitirim™ 5 or 10mg according to SmPC (Summary of Product Characteristics )

Exclusion Criteria:

* History of stress incontinence
* Active urinary tract infection (confirmed by positive urine analysis)
* Symptoms suggestive of severe Bladder Outlet Obstruction (BOO) defined as Qmax<10ml/sc and/or PVR>150ml
* History of known hypersensitivity to solifenacin succinate, oxybutynin hydrochloride, other anti-cholinergics or lactose, to any component of the dosage form or any other allergy, which, in the opinion of the Investigator contraindicates their participation
* Uncontrolled Diabetes Mellitus
* History of drug and/or alcohol abuse at the time of enrolment
* History of acute urinary retention, severe gastrointestinal obstruction (including paralytic ileus or intestinal atony or toxic megacolon or severe ulcerative colitis), myasthenia gravis, uncontrolled narrow glaucoma or swallow anterior chamber or deemed to be at risk of these conditions
* Undergoing haemodialysis or has severe renal impairment or moderate hepatic impairment and who are on treatment with a potent CYP3A4 inhibitor
* History of urogenital tumours which in the opinion of the Investigator precludes their participation in the study
* Likely to participate in another study during study period of 12 weeks from study entry

Min Age: 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified from the Consultants routine clinics and the decision to treat a patient with Vesitirim™ will be made by the treating physician prior to enrolment into this non interventional study
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to visit 2 in Over Active Bladder questionnaire Short Form (OAB-q SF) score | Baseline and 12 weeks
Change from baseline to visit 2 in patient assessment of treatment satisfaction (TS-VAS) | Baseline and 12 weeks

SECONDARY OUTCOMES:
Change from baseline to visit 2 in voiding function assessed by Qmax and PVR | Baseline and 12 weeks
Change from baseline to visit 2 in patient perception of voiding symptoms assessed by: IPSS scores and number of urge incontinence (UUI) episodes per week | Baseline and 12 weeks
Change from baseline to visit 2 in storage symptoms assessed by micturition diary; number of urgency episodes per 24 hours; number of micturition per 24 hours and number of nocturia episodes per 24 hours | Baseline and 12 weeks
Change from baseline to visit 2 in quality of life assessed by IPSS score | Baseline and 12 weeks
Adverse drug reactions- incidence of acute urinary retention and urinary tract infection | Baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Astellas Pharma Co. Ltd (APCL)
Locations (5):
- Ireland (5):
  - Site 2 - Mercy University Hospital, Cork
  - Site: 4 - Tallaght Hospital, Dublin
  - Site: 1 - St James Hopsital, Dublin
  - Site: 5 - Beaumont Hospital, Dublin
  - Site: 3 - Sligo General Hospital, Sligo